CLINICAL TRIAL: NCT06329349
Title: Whole Body and Gut Microbiome Metabolic Flexibility to Predict Lifestyle Intervention Outcomes
Brief Title: Metabolic Flexibility to Predict Lifestyle Interventions Outcomes
Acronym: MEPHISTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government); EXCELES LX22NPO5104, CarDia (Unknown)
Responsible Party: Principal Investigator, Jan Gojda, MD, ass. prof. MD, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK VP57/0/2023
Record Dates: First submitted 2024-03-01; First posted 2024-03-25 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: obesity; metabolic flexibility; metabolomic; exercise; diet
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Intervention Model Description: 2:1 randomized cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Exercise intervention
  Interventions: Other: Exercise; Other: Combined Exercise + Diet
- Control (No Intervention): No intervention.

INTERVENTIONS:
Other: Exercise — 12 weeks, 3 times a week of progressive endurance aerobic exercise (150 to 400kcal AEE per session)
  Arms: Intervention
Other: Combined Exercise + Diet — 12 weeks, 25% caloric reduction, based on PMID: 37069434
  Arms: Intervention

SUMMARY:
Weight loss is a cornerstone of diabetes (T2D) management, yet in clinical practice, its delivery is limited by its perceived burdensome nature and variability in response. Personalization of the interventions to increase their success rate is an unmet clinical need. The proposed project MEPHISTO (Whole body and gut microbiome metabolic flexibility to predict lifestyle intervention outcomes) would aim to identify predictive features related to successful weight loss upon sequential exercise and diet intervention in people living with obesity. To this end, the study aims to conduct a clinical trial where the investigators would implement state-of-the-art physiological phenotyping of metabolic flexibility at the whole-body level and at the level of the gut in persons with obesity before and after exercise and diet + exercise intervention to identify predictive signatures of successful weight loss

DETAILED DESCRIPTION:
Among the influential determinants impacting the efficacy and health outcomes of an intervention is an individual's level of metabolic flexibility (MetFlex). MetFlex denotes the body's capacity to adapt in response to alterations in metabolic demands and nutrient availability. Impaired MetFlex is evident in conditions such as obesity and diabetes, yet it may be ameliorated through lifestyle interventions such as exercise training or caloric restriction similar to improvements in insulin sensitivity. However, MetFlex has not been studied as a potential mechanism associated with successful weight loss. The decline in MetFlex, i.e. the limited cellular/tissue ability to manage excess or deficiency in energy substrates leads to compromised mitochondrial function and excessive lipid accumulation in ectopic tissues, resulting in metabolic disorders such as T2D or metabolic syndrome.

Another potential player predicting an individual's capacity to respond to lifestyle interventions is the gut microbiota (gut microbiome and metabolome, MIME). It was repeatedly shown to be among the most important sources of inter-individual variability when it comes to the development of obesity and responsiveness to dietary intervention The microbiome does not only influence host physiology directly, e.g. through contact with immune cells, but also through the vast array of metabolites produced, i.e. the microbiota-derived metabolome. The composition of the gut microbiota and the microbiota-derived metabolome is largely shaped by the host's diet, as this represents the main source of substances and energy for the microbiota. It is therefore striking that published studies to date have yielded rather inconsistent results regarding dietary interventions to alter gut microbiota composition. The discrepancy can be explained by the large variability of individual microbiomes at the beginning of the intervention, and similarly the baseline MIME signature significantly determines weight loss success.

Here the investigators present a complex project to investigate whether whole body and gut MetFlex can be further explored and used as ex-ante predictors of successful weight loss following exercise and dietary interventions, thus providing proof of concept and paving the way to personalized lifestyle interventions.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30
* age 25-45 years

Exclusion Criteria:

* active cancer
* diabetes (medical history, fasting glycemia >7.6 and/or 2hOGTT glycemia >11.1)
* uncontrolled endocrine diseases
* corticosteroid therapy
* immune-suppressive therapy
* pregnancy
* breastfeeding

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-represented women
Enrollment: 30 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in metabolic flexibility (MetFlex (ΔRQ 200-0)) | 18 months
  change in metabolic flexibility measured as ΔRQ (respiratory quotient) during glucose clamp
Change in insulin sensitivity | 18 months
  change in insulin sensitivity measured as glucose infusion rate (GIR) during glucose clamp

SECONDARY OUTCOMES:
Glucose tolerance relate to primary outcomes changes | 18 months
  fasting/2h oral glucose tolerance test glycemia positively relate to weight loss.
HbA1c relate to primary outcomes changes | 18 months
  HbA1c positively relate to weight loss.
Insulin sensitivity relate to primary outcomes changes | 18 months
  GIR positively relate to weight loss.

OTHER OUTCOMES:
Microbiome composition relate to weight loss: exploratory outcome | 18 months
  Change in microbiome composition in fecal samples upon the intervention is a component of successful weight loss and/or metabolic adaptation
Metabolomic signatures relate to weight loss: exploratory outcome | 18 months
  Change in metabolomic signatures in fecal samples upon the intervention is a component of successful weight loss and/or metabolic adaptation

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gojda, Principal Investigator — Charles University, Czech Republic
Locations (3):
- Czechia (3):
  - University Hospital Kralovske Vinohrady, Prague
  - Third Medical Faculty,Charles University, Prague
  - Faculty of Sports Science, Prague

IPD SHARING:
Plan to Share IPD: No
After anonymization, the data would be shared upon reasonable request.

REFERENCES:
- [Derived] Ludlova M, Koudelkova K, Pallova J, Koudelkova B, Siklova M, Cahova M, Vetrovsky T, Steffl M, Gojda J. Metabolic Flexibility to Predict Lifestyle Interventions Outcomes (MEPHISTO): Protocol for Predictive Validation Study and Randomized Controlled Trial. JMIR Res Protoc. 2025 May 8;14:e67570. doi: 10.2196/67570. PMID 40340957